CLINICAL TRIAL: NCT03680157
Title: Comparing Rater Reliability of Familiar Practitioners to Blinded Coders
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G Welch, Associate Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology) at the Columbia University Medical Center, Developmental Neuroscience, Columbia University
Other Study IDs: AAAS0811
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Child Development; Premature Birth
Keywords: Martha G. Welch; emotional connection; child development; premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine how coders who have seen multiple time points of the same dyad, and are therefore familiar with the case, rate emotional connection using the WECS compared to coders who are blinded to the case's previous time points.

The investigator hypothesizes that the WECS will show external validity: that all coders will have high reliability on their WECS scores, despite exposure to the dyads' past videos by the clinical coders.

DETAILED DESCRIPTION:
The purpose of this study is to determine the external validity of a scale for emotional connection between children and their parents through a retrospective longitudinal study. The Welch Emotional Connection Scale (WECS) is a screen that allows healthcare providers to rate the emotional connection of a mother-child relationship in just a few minutes of observed interaction, and shows preliminary predictive properties when performed in the first year of the child's life. Administration of the WECS involves watching interactions of a child sitting face-to-face on a parent's lap, and scores the interaction on sliding scales in 4 domains. During the WECS development, the Nurture Science Program of Columbia University Medical Center created and coded hours of parent-child interaction videos. This video data set will be used to determine how clinical WECS scores, where raters are familiar with mother-child dyads over time, compare to research WECS scores, where rate-rs are blinded to each case. The WECS scores of clinical coders, who are exposed to the same case at different time points, will be compared to blinded coders who see cases at just one time point. To simulate implementation of the WECS in a clinical setting, two primary care nurse practitioner (PNP) students who are trained in rating emotional connection will view videos to rate the emotional connection of mother-child dyads collected at different time points. To recreate WECS used in a research setting, blinded coders trained in rating emotional connection will rate the emotional connection of the same video data set. Each blinded coder will only view a dyad once, to not be influenced by previous time points of the same subject. The inter-rater reliability of the blinded and clinical coders will be determined. The comparison of inter-rater reliability scores between clinical and blinded coders is the main outcome of this study.

ELIGIBILITY:
Inclusion Criteria:

* Children and their parents who participated in previously conducted studies (AAAD0389)

Exclusion Criteria:

* Children and their parents who had not participated in previously conducted studies (AAAD0389)

Ages: 4 Months to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and their parents who had not participated in previously conducted studies (AAAD0389)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Intra-Class Correlations of Welch Emotional Connection Screen (WECS) Scores | 2018 - 2019
  Blinded Intra-Class Correlations of WECS Scores; Clinical intra-class correlations of WECS Scores. The Welch Emotional Connection Scale (WECS) is an investigational developmental screening tool, developed to rate the quality of the emotional connection that formed between mother and child. The scale is administered in 2-3 minutes by observing a mother and child interact, and requires the rater to critically assess 4 sub-domains of emotional connection. The WECS is scored on intervals of 0.25, with a minimum of 1 (little or no connection) and maximum of 3 (high connection). Separately from these scores, the final portion of the screen determines, "Is the dyad emotionally connected?" and is scored with "No" or "Yes."

CONTACTS AND LOCATIONS:
Overall Officials: Martha Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States